CLINICAL TRIAL: NCT06017349
Title: A Prospective, Multicenter, Open-label, Self-controlled Clinical Trial Protocol to Evaluate the Efficacy and Safety of a Multi-parameter Non-Invasive Glucose Sensors for Measuring Blood Glucose.
Brief Title: To Evaluate the Efficacy and Safety of Multi-parameter Non-Invasive Glucose Sensors for for Blood Glucose Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP-NG -2022-1
Record Dates: First submitted 2023-08-23; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus
Keywords: Blood Glucose Self-Monitoring; Non-invasive glucose meter
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-invasive glucose meter (Experimental): The noninvasive glucose meter was entrained on the finger, Glucose concentration levels were measured by measuring physiological parameters related to metabolic heat and local oxygen supply.
  Interventions: Device: Non-invasive glucose meter
- Accu-Chek Guide blood glucose meter (Active Comparator): Being used for quantitative determination of blood glucose concentration in fresh capillary whole blood taken from fingers.
  Interventions: Device: Accu-Chek Guide
- EKF Biosen C-Line (Active Comparator): Using the hexosyl enzymatic method to detect plasma glucose values
  Interventions: Device: EKF analyzer

INTERVENTIONS:
Device: Non-invasive glucose meter — Blood glucose levels were measured while fasting, after breakfast, and after lunch，Place your index finger into the non-invasive blood glucose meter and wait for the instrument to display the reading.
  Arms: Non-invasive glucose meter
Device: EKF analyzer — Blood glucose levels were measured while fasting, after breakfast, and after lunch，After collecting venous blood and separating plasma, blood glucose detection is performed using the EKF analyzer with the hexokinase method.
  Arms: EKF Biosen C-Line
Device: Accu-Chek Guide — Blood glucose levels were measured while fasting, after breakfast, and after lunch，Use Accu-Chek Guide blood glucose meter to prick the finger and obtain blood for glucose measurement
  Arms: Accu-Chek Guide blood glucose meter

SUMMARY:
This was a prospective, multicenter, open-label, self-controlled study to evaluate the efficacy and safety of multi-parameter non-invasive glucose meters for blood glucose measurement，planned enrollment of 200 patients with type 1 or type 2 diabetes.

Comparing glucose measurements from the Non-Invasive Glucose monitoring system to venous blood glucose or fingertip blood glucose to evaluate System accuracy capability.

DETAILED DESCRIPTION:
At the same time, blood glucose was measured by non-invasive blood glucose meter, Accu-Chek Guide blood glucose meter and EKF Biosen C-Line. Eight groups of blood glucose values were collected from each subject during fasting, after breakfast and after lunch.After the end of blood glucose measurement, the data were recorded, including adverse events and device defects during the test. The subjects were required to stay in the examination room for 5-10 minutes, during which they completed the product use evaluation questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diabetes (type 1 or type 2 );
* Participants who could understand the purpose of the trial and signed the informed consent form.

Exclusion Criteria:

* Conditions that prevent good contact between the measuring finger and the sensor, resulting in unmeasured conditions, such as hand disability, scar, swelling of the finger, etc.
* Diseases that affect the accuracy of hand measurement, such as Parkinson's disease, upper limb chronic arterial occlusive disease, Raynaud's syndrome, hand or arm trauma surgery, upper limb arteriovenous fistula, etc.
* Fever (axillary temperature >37.3℃) and severe dehydration during screening;
* Diabetic ketoacidosis, hyperglycemic hyperosmolar status within 6 months before signing the informed consent;
* Those who were in serious illness within 1 month before signing the informed consent, such as shock, heart failure, respiratory failure, severe liver and kidney dysfunction, etc.
* Those suffering from mental illness, lack of self-control or unable to express their personal willingness clearly;
* Participants who participated in other drug or device clinical trials within 2 weeks before signing the informed consent (except those who failed in screening);
* Other persons deemed by the investigator to be ineligible for clinical trial participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
The results were analyzed by consensus error grid (CEG) | After 2 days of blood glucose measurements
  The proportion of the results lie within zone A and zone B of the consensus error grid (CEG)

SECONDARY OUTCOMES:
Mean Absolute Relative Difference (MARD) | The day after the blood glucose measurement
  It is calculated by taking the absolute difference between the two values, dividing it by their average. A smaller MARD value indicates a smaller relative difference between the two values, indicating higher consistency between them.
The 20/20% agreement rates | The day after the blood glucose measurement
  the proportion of Non-invasive blood glucose values that were within 20% of paired reference blood glucose values >80 or 20 mg/dL of reference blood glucose values ≤100 mg/dL
Accessibility evaluation Questionnaire for non-invasive glucose meter | The day after the blood glucose measurement
  The questionnaire covers the subjects' self-monitoring of blood glucose status, their awareness and expectations of non-invasive testing, as well as their subjective feelings after using a non-invasive blood glucose meter.

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China